CLINICAL TRIAL: NCT05991687
Title: Methods for Effective Disposal of Surplus Analgesics to Facilitate Elimination
Acronym: MEDSAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Mark Bicket, MD, PhD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00236974; E20233700-001 (Other Grant/Funding Number: Michigan Department of Health and Human Services)
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Analgesics, Opioids
Keywords: Opioids; Drug disposal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-home (Active Comparator)
  Interventions: Other: In-home drug disposal pouch
- Mail-in (Active Comparator)
  Interventions: Other: Mail-in prepaid envelope

INTERVENTIONS:
Other: In-home drug disposal pouch — Will receive a drug disposal pouch to inactivate leftover prescription opioids for disposal after surgery.
  Arms: In-home
Other: Mail-in prepaid envelope — Will receive a prepaid envelope to mail leftover prescription opioids for disposal after surgery
  Arms: Mail-in

SUMMARY:
The primary objective is to evaluate the difference in outcomes for mail-in vs. in-home disposal methods for leftover prescription opioids after discharge from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated to be prescribed and use an opioid medication to treat acute pain after elective outpatient surgery
* Opioid-naive

Exclusion Criteria:

* Inability to receive email and/or phone calls for follow up assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Use of assigned disposal method | 2 weeks after surgery
  Among patients who have leftover opioids, patient report of the use of their assigned mail-in or in-home method of disposal by 2 weeks after surgery.

SECONDARY OUTCOMES:
Use of safe disposal method | 2 weeks after surgery
  Patient-reported use of a method for disposal of leftover opioids that includes mail-in, in-home, pharmacy drop off, or flushing down the toilet by
Use of any disposal method | 2 weeks after surgery
  Patient-reported use of any method to dispose of leftover opioids, that includes assigned methods, safe methods, and other methods such as placing in the trash
Feasibility of Intervention Measure (FIM) | 2 weeks after surgery
Acceptability of Intervention Measure (AIM) | 2 weeks after surgery
Patient-Reported Satisfaction with Use of Disposal Method (study derived question) | 2 weeks after surgery
  Patient report of overall satisfaction with use of the assigned disposal method, on a 0 (worst) to 10 (best) numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bicket, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No